CLINICAL TRIAL: NCT05056584
Title: The Role of the Kidneys and Liver in the Elimination of Glucagon An Evaluation of the Metabolic Clearance Rate of Glucagon in Patients With End-stage Renal Disease and Patients With Liver Cirrhosis
Brief Title: The Role of the Kidneys and Liver in the Elimination of Glucagon
Acronym: MCR_EndCir
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: The Novo Nordisk Foundation Center for Basic Metabolic Research (Other)
Responsible Party: Principal Investigator, Magnus Frederik Gluud Grøndahl, Principal investigator, Medical Doctor, University Hospital, Gentofte, Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-16043802
Record Dates: First submitted 2020-11-09; First posted 2021-09-24 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Chronic Kidney Diseases; Liver Cirrhosis; Hyperglucagonemia
Keywords: Metabolic clearance rate; Glucagon pharmacodynamics; Glucagon pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency, Chronic; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy control subjects (Experimental): Healthy control subjects, matched for age, sex and BMI
  Interventions: Biological: Glucagon infusion; Biological: Primed tracer infusion
- Patients with End-stage Renal Disease (Experimental): Patients with hemodialysis-treated ESRD.
  Interventions: Biological: Glucagon infusion; Biological: Primed tracer infusion
- Patients with liver cirrhosis (Experimental): Patients with Child-Pugh A or B Cirrhosis
  Interventions: Biological: Glucagon infusion; Biological: Primed tracer infusion

INTERVENTIONS:
Biological: Glucagon infusion — One hour glucagon-clamp followed by one hour of blood sampling
Biological: Primed tracer infusion — Infusion of primed isotopically labelled glucose, amino acids and lipids. From 2 hours prior to glucagon infusion and throughout the test day,

SUMMARY:
The study aims to evaluate the kinetics and effect of glucagon in patients with chronic kidney disease and liver cirrhosis and matched healthy subjects, respectively.

DETAILED DESCRIPTION:
In the present project the investigators wish to identify whether the effect, elimination and degradation of glucagon differ between healthy control subjects and patients with Chronic Kidney Disease (CKD) and liver cirrhosis, respectively. By performing glucagon infusions on healthy control subjects and matched subjects with either limited renal and hepatic function, the contribution of both organs to the metabolic clearance rate (MCR) of glucagon can be tested. A primed infusion of stable isotopic labelled tracers will allow the researchers to investigate the effects of the glucagon infusion on the glucose, lipid and amino acid metabolism.

The quantification of the MCR of glucagon will be accompanied by a range of pharmacodynamic measures in order to substantiate whether a potentially altered glucagon MCR inflicts pharmacodynamic changes of glucagon, which could contribute to the pathophysiology of CKD and liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

The CKD group

* Men/women between 18 and 75 years of age
* CKD stage 4 or 5
* Normal liver function (alanine aminotransferase (ALAT), aspartate aminotransferase (ASAT), albumin and coagulation factor II, VII and X (INR) within normal range,
* Informed consent

The cirrhosis group

* Men/women between 18 and 75 years of age
* Verified diagnosis of cirrhosis - Child-Pugh Score of 5-12
* Normal kidney function (estimated glomerular filtration rate (eGFR) above 60 ml/min/1.73m2 and absence of proteinuria)
* Informed consent

The control group

* Men/women between 18 and 75 years of age
* Normal kidney function (estimated glomerular filtration rate (eGFR) above 60 ml/min/1.73m2 and absence of proteinuria)(plasma creatinine ≤105 micromol/L (µM) for men and ≤90 µM for women)
* Normal liver function (alanine aminotransferase (ALAT), aspartate aminotransferase (ASAT), albumin and coagulation factor II, VII and X (INR) within normal range
* Informed consent

Exclusion Criteria:

All groups

* Diagnosis of diabetes and/or HbA1c ≥43 mmol/mol and/or fasting plasma glucose ≥6 mmol/l.
* Previous kidney transplantation with remaining kidney graft
* Present treatment with oral glucocorticoids
* Polycystic kidney disease
* Pregnancy or breastfeeding
* Inflammatory bowel disease
* Surgical procedure within the last 3 months
* Haemoglobin < 6 mmol/l (women) or < 7 mmol/l (men)
* First-degree relatives with diabetes
* Any condition that the investigators feel would interfere with trial participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Metabolic clearance rate of glucagon | t = 50 minutes
  Glucagon plasma concentration steady state glucagon concentrations

SECONDARY OUTCOMES:
Glucagon pharmacokinetic 1 | -120, -90, -60, -30, -15, 0, 5, 10, 20, 50, 55, 60, 62, 64, 66, 68, 70, 75, 80, 85, 90, 120 minutes
  Elimination half-life
Glucagon pharmacokinetic 2 | -120, -90, -60, -30, -15, 0, 5, 10, 20, 50, 55, 60, 62, 64, 66, 68, 70, 75, 80, 85, 90, 120 minutes
  volume of distribution of Glucagon
Glucagon pharmacodynamic - amino acids | -120, -90, -60, -30, -15, 0, 5, 10, 20, 50, 55, 60, 62, 64, 66, 68, 70, 75, 80, 85, 90, 120 minutes
  Effect of glucagon on amino acid plasma levels before, during and after infusion
Glucagon pharmacodynamic - glucose | -120, -90, -60, -30, -15, 0, 5, 10, 20, 50, 55, 60, 62, 64, 66, 68, 70, 75, 80, 85, 90, 120 minutes
  Effect of glucagon on plasma glucose levels before, during and after infusion
Tracers | -120, -90, -60, -30, -15, 0, 5, 10, 20, 50, 55, 60, 62, 64, 66, 68, 70, 75, 80, 85, 90, 120
  Tracer-to-tracee ratio of labelled isotopes
Insulin | -120, -90, -60, -30, -15, 0, 5, 10, 20, 50, 55, 60, 62, 64, 66, 68, 70, 75, 80, 85, 90, 120 minutes
  Excursions of plasma concentrations of insulin
Glucagon-like peptide 1 | -120, -90, -60, -30, -15, 0, 5, 10, 20, 50, 55, 60, 62, 64, 66, 68, 70, 75, 80, 85, 90, 120 minutes
  Excursions of plasma concentrations of GLP-1
Lipid metabolism | -120, -90, -60, -30, -15, 0, 5, 10, 20, 50, 55, 60, 62, 64, 66, 68, 70, 75, 80, 85, 90, 120 minutes
  Effect of glucagon on lipid metabolism, through lipidomics
Vital parameter 1 | -120, -30, 0, 60, 120 minutes
  Systolic blood pressure
Vital parameter 2 | -120, -30, 0, 60, 120 minutes
  Diastolic blood pressure
Vital parameter 3 | -120, -30, 0, 60, 120 minutes
  Heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, PhD, Study Director — Center for Metabolic Research, Gentofte Hospital; Magnus FG Grøndahl, MD, Principal Investigator — Center for Metabolic Research, Gentofte Hospital
Locations (1):
- Center for Clinical Metabolic Research, Department of Medicine, Gentofte Hospital, Hellerup, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No